CLINICAL TRIAL: NCT03896802
Title: Hemodynamic Effects of PEEP in Patients With ARDS
Brief Title: Hemodynamic Effects of PEEP in ARDS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Davide Chiumello, Director of Intensive Care, University of Milan
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: ARDS-HEMO
Record Dates: First submitted 2019-03-28; First posted 2019-04-01 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Acute Respiratory Distress Syndrome; Mechanical Ventilation; ARDS, Human
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low PEEP (Experimental): PEEP 5 cmH2O
  Interventions: Procedure: Physiological assesment
- High PEEP (Experimental): PEEP 15 cmH2O
  Interventions: Procedure: Physiological assesment

INTERVENTIONS:
Procedure: Physiological assesment — 1. Arterial and mixed venous blood gas analysis.
  2. Alveolar and physiologic dead space via volumetric capnometry, as well as carbon dioxide (CO2) production, end-tidal CO2 and mixed expired CO2
  3. Respiratory system (Crs), chest wall (Ccw) and lung (Cl) compliance measurement via an end-inspiratory and end-expiratory pause.
  4. Arterial blood pressure, central venous pressure (CVP), heart rate, cardiac output through the arterial pulse contour and transpulmonary thermodilution methods (PiCCO technology). Global end-diastolic volume, Intra-thoracic blood volume, Extravascular lung water will also be assessed. Respiratory hold maneuvers (at PEEP, and +10, +15 and +20 cmH2O) will be performed and CVP and cardiac output will be measured in the last 3 s of the 12 s inspiratory hold. Venous return curve will constructed and the zero-flow pressure recorded as the mean systemic filling pressure.
  5. Urine flow in 1h and determination of the fractional excretion of sodium and creatinine.

SUMMARY:
The purpose of this study is to assess the effect of different levels of PEEP on the cardiocirculatory system in patients affected by the acute respiratory distress syndrome (ARDS)

DETAILED DESCRIPTION:
Introduction

Acute respiratory distress syndrome (ARDS) is a clinical syndrome defined by the association of an acute onset of hypoxaemia and bilateral pulmonary infiltrates following a trigger insult; it is characterized by inflammation of the pulmonary tissue, with subsequent development of non-cardiogenic edema. The extent of edema may be such that the weight of the lung may increase up to 2-3 times its original weight. As a consequence, the lung tends to collapse on itself, more so in the dependent areas, i.e. the posterior/dorsal areas when the patient in lying supine, with the consequent development of zones of atelectasis.

These areas, when perfused, are the main cause for the development of the severe form of hypoxemia commonly seen in this condition. Hypoxemia, if severe enough, may bring by itself to the death of the patient. It has to be noted that, despite the advances in the management of critically ill patients, mortality attributable to ARDS currently is about 50%, with a range between 30-70%.

The use of positive end-expiratory pressure (PEEP) has been reported ever since the first description of the syndrome, as a tool to manage and correct hypoxemia. PEEP has thus been used for 40 years, and is an essential part of the management of the syndrome. While the effectiveness of PEEP in improving the oxygenation of the wide part of critically ill patients with ARDS it is out of doubt, its efficacy with respect to outcomes such as mortality has not, so far, been demonstrated. The question is then still open with regards to the setting of an optimal level of PEEP in ARDS.

Frequently, ARDS is associated with the development of hemodynamic instability and shock, to the extent that up to 2/3 of patients suffering from the syndrome require the infusion of catecholamines or show signs of hypoperfusion; circulatory failure seems to be the factor more strongly associated to mortality in these patients, and the strength of the association is higher compared to that of the degree of hypoxemia. In ARDS shock is secondary to three main factors: 1) acute cor pulmonale due to pulmonary hypertension secondary to microvascular occlusion by thrombi or arteriolar remodeling and/or hypoxic pulmonary vasoconstriction; 2) the deleterious hemodynamic effects of mechanical ventilation, especially on right cardiac function; and 3) the possible development of septic myocardial depression.

Acute kidney injury (AKI) is common in critically ill patients and it is associated with poor outcomes. An increasing body of evidence points to the existence of deleterious interactions between kidney and lung dysfunctions in a vicious cross-talk. Several studies seem to suggest that mechanical ventilation and ARDS may have adverse effects on kidney function via three main mechanisms: 1) positive-pressure ventilation may lead to a reduction in cardiac output and an increase central venous pressure, thereby diminishing renal blood flow, free water clearance, and the glomerular filtration rate; 2) changes in arterial blood oxygen (O2) or carbon dioxide (CO2) may influence renal vascular resistance, renal perfusion, or diuresis; and, finally, 3) emerging data suggest that ventilator-induced lung injury may not only affect the lung, but may also lead to further systemic inflammation via the systemic release of inflammatory cytokines.

Indeed, the hemodynamic effect of PEEP depends on how much of the positive pressure applied to the alveoli is transmitted to the mediastinal structures (heart and big vessels), and the effect on renal function depends on how much this interferes with renal hemodynamic. The transmission of airway pressure, in turn, depends on the mechanical characteristics of the lung and the chest wall, which are known to be variably and unpredictably affected in ARDS.

The main question of this research project deals with the hemodynamic impact of PEEP in patients with ARDS, in terms of effects on the cardiocirculatory system.

Rationale

Hemodynamic effects of mechanical ventilation The hemodynamic effects of mechanical ventilation are mainly secondary to cyclic oscillations in pleural pressure (Ppl) and transpulmonary pressure (Ptp). Variations in pleural pressure mainly interfere with inflow of blood into the right ventricle, and with ejection of blood from the left ventricle. On the other side, variations in transpulmonary pressure mainly affect the inflow of blood into the left ventricle and ejection of blood from the right ventricle. While the large vessels of systemic circulation are surrounded by the constant atmospheric pressure, central vessels of the pulmonary circulation are surrounded by pleural pressure, which in turn may significantly vary compared to atmospheric pressure during the whole respiratory cycle. Positive-pressure mechanical ventilation exerts an effect which is opposed to the physiologic inspiratory negativisation of pleural pressure. Indeed, the increase in pleural pressure secondary to positive airway pressure reduces left ventricular afterload, while at the same time it reduces right ventricular preload. Since the normal pressure gradient which drives blood from periphery to the right heart lies in the range of 4-8 mmHg, even small increases in pleural pressure may have a significant impact on venous return. Moreover, the presence of PEEP has a hemodynamic effect during the whole respiratory cycle. As a rule of thumb, it is generally estimated that up to about 50% of the variation in airway pressure is transmitted as a variation in pleural pressure in patients with normally functioning lungs. This effect is however likely reduced in case of an increased lung elastance (i.e. the presence of stiff lungs, as in patients with ARDS), given that a reduced amount of airway pressure is transmitted at the pleural level. However, this depends on the ratio between lung elastance and respiratory system elastance, which may vary widely in ARDS. Moreover, as the right ventricle generally displays a high level of compliance despite a limited myocardial thickness and a reduced contractile force, this may be more affected from increments in afterload rather than by variations in preload.

On the other side, the increase in mean airway pressure as a consequence of the application of PEEP leads to an increase in the size of the lung (increase in end-expiratory lung volume), mainly through the recruitment of previously closed and derecruited zones. However, the application of PEEP may also lead to overdistention of already open and ventilated pulmonary units, leading to a certain degree of vascular occlusion of the critical closing pressure of those vessels is reached and overcome (as in the case of West zones I and II, in which alveolar pressure in higher than arterial and venous pulmonary pressure, respectively).

The hemodynamic effect of PEEP might then be different, as a function of the amount of pulmonary units that can be recruited. In conclusion, the knowledge of the effect on the cardiocirculatory system of the application of a high or low level of PEEP may require the measure or at least an estimate of the potential for lung recruitment.

Measurement and estimate of the potential for lung recruitment The gold standard for the measurement of the potential for lung recruitment is represented by pulmonary CT scan. This technique has been used together with quantitative analysis of regional and global lung aeration by our group since 1987 for the analysis of parenchymal response to PEEP in patients with ARDS. An estimate of the potential for lung recruitment may be inferred at the bedside by the assessment of the effect of PEEP on the level of oxygenation, physiologic dead-space and partitioned lung compliance, to be able to differentiate recruitment from overdistention.

Main hypothesis The main hypothesis behind the present research project is that critically ill patients with ARDS and an elevated potential for lung recruitment will be less affected by the hemodynamic effects of PEEP than patients with a lower potential for lung recruitment. If this hypothesis was to be confirmed, the application of PEEP would be less troublesome, at least for the concerns for the hemodynamic compromise, in patients with ARDS and a higher potential for lung recruitment. This issue has so far never been investigated, and the present research might significantly extend our knowledge on the topic.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged 18 or older and with a recent (<48h) diagnosis of ARDS, undergoing invasive mechanical ventilation and in whom, due to the hemodynamic instability, cardiac output monitoring with an Arterial pulse contour analysis and transpulmonary thermodilution system (PiCCO technology, Pulsion Medical Systems, Germany) will be considered necessary, will be considered for enrolment.

Exclusion Criteria:

* Patients with barotrauma and with clinical evidence of intrinsic PEEP will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Cardiac Output | Study 1 day
  Cardiac output (in l/min) will be measured by transpulmonary thermodilution and arterial pulse contour analysis

SECONDARY OUTCOMES:
Transmural central venous pressure | Study 1 day
  Measured and CVP minus esophageal pressure
Mean systemic filling pressure | Study 1 day
  Measured with the respiratory hold method

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale San Paolo - Polo Universitario, ASST Santi Paolo e Carlo, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: No